CLINICAL TRIAL: NCT03629925
Title: A Randomized, Double-Blind, Phase III Study to Compare the Efficacy and Safety of Sintilimab (IBI308) in Combination With Gemcitabine and Platinum-Based Chemotherapy vs. Placebo in Combination With Gemcitabine and Platinum-Based Chemotherapy as First-Line Treatment for Patients With Advanced or Metastatic Squamous Non-Small-Cell Lung Cancer (NSCLC) (ORIENT-12)
Brief Title: Sintilimab in Combination With Gemcitabine and Platinum-Based Chemotherapy as First-Line Therapy for Advanced or Metastatic Squamous NSCLC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIBI308C303
Record Dates: First submitted 2018-08-09; First posted 2018-08-14 (Actual); Results first posted 2021-04-01 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Squamous NSCLC
MeSH Terms: interventions — sintilimab; Gemcitabine; Cisplatin; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sintilimab+ gemcitabine plus platinum (Experimental): Sintilimab combination arm: Sintilimab in combination with gemcitabine plus cisplatin or carboplatin
  Interventions: Drug: Sintilimab; Drug: Gemcitabine; Drug: Cisplatin; Drug: Carboplatin
- Placebo+gemcitabine plus platinum (Placebo Comparator): Placebo combination arm: Placebo in combination with gemcitabine plus cisplatin or carboplatin
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Drug: Placebo; Drug: Carboplatin

INTERVENTIONS:
Drug: Sintilimab — 200mg, Q3W, day1, I.V.; consecutive cycles
  Other Names: IBI308
  Arms: Sintilimab+ gemcitabine plus platinum
Drug: Gemcitabine — 1000mg/m^2, Q3W, day 1and 8, I.V.; first 4 or 6 consecutive cycles.
Drug: Cisplatin — 75 mg/m^2, Q3W, day1, I.V.; first 4 or 6 consecutive cycles.
Drug: Placebo — NA, Q3W, day1, I.V.; consecutive cycles
  Arms: Placebo+gemcitabine plus platinum
Drug: Carboplatin — AUC 5mg/ml/min, Q3W, day1, I.V.; first 4 or 6 consecutive cycles.

SUMMARY:
Efficacy and Safety Evaluation of IBI308 in Patients with Advanced or Recurrent Squamous NSCLC

DETAILED DESCRIPTION:
The anti-tumor activity of anti-PD-1 therapy in previously untreated Chinese squamous NSCLC patients will be investigated in this clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must sign written ICF prior tothe implementation of any procedures related to the study;
2. Aged ≥ 18 years and ≤ 75 years;
3. With a life expectancy of more than 3 months;
4. With at least one measurable lesion confirmed by the investigator according to RECIST v1.1.

   Measurable lesions locatedin the field of previous radiotherapy or locoregional therapy canbe selected as target lesions if PD is confirmed;
5. Participants with histologically or cytologically confirmed locally advanced (stage IIIB/IIIC) who are ineligible for radical surgery or concurrent chemoradiotherapy, metastatic (stage IV)or recurrent squamous NSCLC based on the "8th Edition of the TNM Classification for LungCancer" issued by the International Association for the Study of Lung Cancer and the American Joint Committee on Cancer Classification;
6. With an ECOG PS score of 0 or 1;
7. Have not received any prior systemic anti-tumor therapy for advanced/metastatic disease; for participants who have received prior platinum-based adjuvant chemotherapy/radiotherapy,neoadjuvant chemotherapy/radiotherapy, or radical chemoradiotherapy, they are eligible for the study if PD occurs at > 6 months after the last treatment;
8. With adequate hematologic function, defined as ANC ≥ 1.5 × 10^9/L, platelet count ≥ 100 × 10^9/L, and hemoglobin ≥ 90 g/L (noblood transfusion history within 7 days);
9. Adequate hepatic function, defined as TBIL ≤ 1.5 × ULN and AST as well as ALT ≤ 2.5 × ULN for all participants, or AST and ALT ≤ 5 × ULN for participants with liver metastasis;
10. Adequate renal function, defined as CCr ≥ 50 mL/min (Cockcroft-Gault formula);
11. Adequate coagulation function, defined as INR or PT ≤ 1.5 × ULN; for the participant who is receiving anticoagulant therapy, INR or PT within the proposed scope of the anticoagulantmedication is acceptable;
12. Female participants of childbearing age should be tested negative for urine or serum pregnancy within 3 days before the first dose of the study treatments. A blood pregnancy testis required if the urine pregnancy test is inconclusive;
13. For male and female participants with conception potential, highly effective contraception measures (failure rate < 1% per year) should be taken until at least 180 days afterdiscontinuation of the study treatment;

Note: Abstinence is acceptable as a method of contraception if it is the usual lifestyle and preferred method of contraception for the participant.

Exclusion Criteria:

1. Histological type of nonsquamousNSCLC. The dominant cell morphology must be identified for mixed cell type (participants with squamous cell carcinoma components > 50% can beenrolled); participants with small cell carcinoma, neuroendocrine carcinoma, and sarcoma components cannot be included;
2. Participants with known EGFR-sensitive mutations or ALK rearrangement;
3. Currently participating in an interventional clinical study, or treated with another study drug therapy or investigational device therapy within 4 weeks before the first dose;
4. Previously received the following therapies: anti-PD-1, anti-PD-L1, or anti-PD-L2 agents or agents targeting another stimulation or synergistically inhibiting TCR (e.g., CTLA-4, OX-40,and CD137);
5. Received proprietary Chinese medicines with anti-tumor indications or immunomodulators (thymosin, interferon, interleukin, etc.) within 2 weeks prior to the first dose, or received a major surgery within 3 weeks prior to the first dose;
6. With active hemoptysis, active diverticulitis, abdominal abscess, gastrointestinal obstruction, and peritoneal metastases requiring clinical intervention;
7. Have undergone solid organ transplantation or hematologic transplantation;
8. With clinically uncontrolled pleural effusion/ascites (participants who do not need effusion drainage or have no significant increase in effusion within 3 days after stopping drainage canbe enrolled);
9. With a tumor compressing the surrounding important organs (such as esophagus) with relevant symptoms, compressing the superior vena cava, or invading the mediastinal great vessels,heart, etc.;
10. With Class III-IV congestive cardiac failure (based on New York Heart Association Classification) or poorly controlled and clinically significant arrhythmia;
11. With any arterial thrombosis, embolism, or ischemia within 6 months prior to enrollment, such as myocardial infarction, unstable angina, cerebrovascular accident, and transient ischemicattack. With a history of deep venous thrombosis, pulmonary embolism, or any other seriousthromboembolic events within 3 months priorto enrollment (implantable port or catheter-related thrombosis, or superficial venous thrombosis is not considered as "serious"thromboembolism);
12. With known allergy to the active ingredients and/or any excipient of sintilimab , gemcitabine, cisplatin, orcarboplatin;
13. With active autoimmune disease requiring systemic treatment (e.g., use of disease-modifying drugs, corticosteroids, or immunosuppressive agents) within 2 years before the first dose.Replacement therapy (e.g., thyroxine, insulin, or physiologic doses of corticosteroids foradrenal or pituitary insufficiency) is not considered systemic;
14. Participants requiring long-term systemic use of corticosteroids. Participants requiring intermittent use of bronchodilators, inhaled corticosteroids, or localinjection ofcorticosteroids for COPD or asthma can be included in the study;
15. Full recovery (i.e., ≤ Grade 1 or reaching the baseline, excluding asthenia or alopecia) from toxicity and/or complications caused by any intervention has not achieved before thestart oftreatment;
16. Diagnosed with other malignant tumors within 5 years before the first dose, excluding radically cured cutaneous basal cell carcinoma, cutaneous squamous cell carcinoma, and/orradically resected carcinoma in situ. For other malignant tumors or lung cancer diagnosedmore than 5 years before the first dose, pathological or cytological diagnosis should beperformed for recurrent and metastatic lesions;
17. Symptomatic CNS metastasis. Participants with asymptomatic brain metastases or with stable symptoms after treatment of brain metastases are allowed to participate in this study as longas meeting all of the following criteria: presence of measurable lesions outside the CNS;absence of metastases in midbrain, pons, cerebellum, meninges, medulla oblongata, or spinalcord; maintain clinical stable condition for at least 2 weeks; discontinue hormone therapy 14 days prior to the first dose of the study treatments;
18. With a history of non-infectious pneumonia requiring corticosteroid therapy within 1year prior to the first dose or with non-infectious pneumonia at present;
19. With an active infection requiring treatment or have used systemic anti-infective drugs within one week prior to the first dose;
20. With known psychiatric disorder or substance abuse that could affect the compliance with study requirements;
21. Known history of HIV infection (i.e. HIV 1/2 antibody positive), known syphilis infection (syphilis antibody positive), or active tuberculosis;
22. With untreated active hepatitis B;

    Note: Participants with hepatitis B who meet the following criteria are also eligible forinclusion:

    HBV viral load must be less than 1000 copies/mL (200 IU/mL) or below LLD prior to thefirst dose, and participants should receive anti-HBV treatment to avoid virus reactivation throughout the therapeutic phase of the study; For participants with HBcAb (+), HBsAg (-), HBsAb (-), and HBV load (-), close monitoring is required instead of prophylactic anti-HBV treatment to avoid virus reactivation;
23. Participants with active HCV infection (HCV antibody positive and HCV-RNA level above the LLD);
24. Have received live vaccines within 30 days prior to the first dose; Note: Seasonal inactivated influenza virus vaccines for injection are allowed, while liveattenuated influenza vaccines forintranasal use are not acceptable;
25. With any medical history, disease, treatment, or laboratory abnormal finding that would interfere with the study results or prevent the participant from participating in the whole study,or the investigator believes that participation in this study is not in the best interest of theparticipant;
26. With local or systemic diseases not attributing to malignancy, or with cancer-related secondary diseases, which would result in a high medical risk and/or uncertainty in survivalevaluation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Jiang M, Sun J, Hu C, Wu L, Fan Y, Wang Z, Liu L, Wu C, Wu F, Gao G, Li F, Wang L, Li X, Cheng L, Peng B, Zhou H, Zhou C. A tumor cornification and immune-infiltration-based scheme for anti-PD-1 plus chemotherapy response in advanced squamous cell lung carcinoma. Med. 2025 Feb 14;6(2):100516. doi: 10.1016/j.medj.2024.09.005. Epub 2024 Oct 11. PMID 39395411
- [Derived] Zhou C, Wu L, Fan Y, Wang Z, Liu L, Chen G, Zhang L, Huang D, Cang S, Yang Z, Zhou J, Zhou C, Li B, Li J, Fan M, Cui J, Li Y, Zhao H, Fang J, Xue J, Hu C, Sun P, Du Y, Zhou H, Wang S, Zhang W. Sintilimab Plus Platinum and Gemcitabine as First-Line Treatment for Advanced or Metastatic Squamous NSCLC: Results From a Randomized, Double-Blind, Phase 3 Trial (ORIENT-12). J Thorac Oncol. 2021 Sep;16(9):1501-1511. doi: 10.1016/j.jtho.2021.04.011. Epub 2021 May 25. PMID 34048947

RESULTS

PARTICIPANT FLOW:
Recruitment Details: primary analysis data cutoff date: 15 October 2019; updated analysis data cutoff date: 25 March 2020
Groups:
- Sintilimab+ Gemcitabine Plus Platinum: Sintilimab 200mg IV, Gemcitabine 1.0 g/m^2 IV and Cisplatin 75 mg/m^2 or Carboplatin AUC 5 mg/ml/min IV Q3W.
- Placebo+Gemcitabine Plus Platinum: Placebo IV, Gemcitabine 1.0 g/m^2 IV and Cisplatin 75 mg/m^2 or Carboplatin AUC 5 mg/ml/min IV Q3W.
Period: Overall Study
Arm/Group | Sintilimab+ Gemcitabine Plus Platinum | Placebo+Gemcitabine Plus Platinum
Started | 179 | 178
Completed | 0 | 0
Not Completed | 179 | 178

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sintilimab+ Gemcitabine Plus Platinum | Placebo+Gemcitabine Plus Platinum | Total
Number analyzed (Participants) | 179 | 178 | 357
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.9 (7.47) | 61.0 (7.85) | 61.5 (7.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 30
  Male | 163 | 164 | 327
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 179 | 178 | 357
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 179 | 178 | 357
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 179 | 178 | 357

OUTCOME MEASURES:

1. Primary Outcome: PFS(Progression Free Survival)
Description: PFS was defined as the time from randomization to the first documented PD or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. PFS according to RECIST 1.1 as assessed by BIRRC was reported for each arm.
Time Frame: Through Database Cutoff Date of 25 March 2020 (up to approximately 18 months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sintilimab+ Gemcitabine Plus Platinum | Placebo+Gemcitabine Plus Platinum
Number analyzed (Participants) | 179 | 178
months | 5.5 [4.9 to 6.8] | 4.9 [4.8 to 5.0]

2. Secondary Outcome: OS (Overall Survival)
Description: OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were to be censored at the date of the last follow-up. OS was reported for each arm.
Time Frame: Through Database Cutoff Date of 15 October 2019 (up to approximately 13 months)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sintilimab+ Gemcitabine Plus Platinum | Placebo+Gemcitabine Plus Platinum
Number analyzed (Participants) | 179 | 178
Months | NA [NA to NA] — Median OS and upper and lower limit of 95%CI not reached due to insufficient number of participants with events | NA [NA to NA] — Median OS and upper and lower limit of 95%CI not reached due to insufficient number of participants with events

3. Secondary Outcome: ORR(Objective Response Rate)
Description: ORR was defined as the percentage of participants in the analysis population who had a confirmed Complete Response (CR: disappearance of all lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters [SOD] of target lesions, taking as reference the baseline SOD) according to RECIST 1.1. The percentage of participants who experienced a confirmed CR or PR according to RECIST 1.1 as assessed by BIRRC was reported as the ORR for each arm.
Time Frame: Through Database Cutoff Date of 25 March 2020 (up to approximately 18 months)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Sintilimab+ Gemcitabine Plus Platinum | Placebo+Gemcitabine Plus Platinum
Number analyzed (Participants) | 179 | 178
Percentage of Participants | 44.7 [37.27 to 52.29] | 35.4 [28.38 to 42.90]

4. Secondary Outcome: TTR (Time to Response)
Description: TTR was defined as the time of participants from the first treatment administration to the first incidence of a confirmed CR (disappearance of all lesions) or PR (at least a 30% decrease in the sum of diameters [SOD] of target lesions, taking as reference the baseline SOD) according to RECIST 1.1. The time from first treatment administration to the first incidence of treatment response was reported as the TTR for each arm.
Time Frame: Through Database Cutoff Date of 25 March 2020 (up to approximately 18 months)
Measure: Median (Full Range); unit: Months
Arm/Group | Sintilimab+ Gemcitabine Plus Platinum | Placebo+Gemcitabine Plus Platinum
Number analyzed (Participants) | 80 | 63
Months | 1.41 [1.2 to 11.1] | 1.41 [1.2 to 2.9]

5. Secondary Outcome: DCR (Disease Control Rate)
Description: DCR was defined as the percentage of participants who had a CR (disappearance of all target lesions), PR (at least a 30% decrease in the sum of diameters of target lesions), or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered PD]). The percentage of participants who experienced a confirmed CR, PR, or SD according to RECIST 1.1 as assessed by BIRRC was reported as the DCR for each arm.
Time Frame: Through Database Cutoff Date of 25 March 2020 (up to approximately 18 months)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Sintilimab+ Gemcitabine Plus Platinum | Placebo+Gemcitabine Plus Platinum
Number analyzed (Participants) | 179 | 178
Percentage of Participants | 86.0 [80.08 to 90.75] | 80.3 [73.73 to 85.91]

6. Secondary Outcome: DOR (Duration of Response)
Description: For participants who demonstrated a confirmed CR (disappearance of all target lesions) or PR (At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR was defined as the time from first documented evidence of a CR or PR until progressive disease (PD) or death. DOR for participants who had not progressed or died at the time of analysis was censored at the date of their last tumor assessment. Per RECIST 1.1, PD was defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered PD. DOR assessments were based on BIRRC assessment. The DOR according to RECIST 1.1 for all participants who experienced a confirmed CR or PR was reported for each arm.
Time Frame: Through Database Cutoff Date of 25 March 2020 (up to approximately 18 months)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sintilimab+ Gemcitabine Plus Platinum | Placebo+Gemcitabine Plus Platinum
Number analyzed (Participants) | 80 | 63
Months | 6.05 [4.73 to 9.63] | 5.06 [3.71 to 5.55]

ADVERSE EVENTS:
Time Frame: Through database cutoff date of 25 March 2020 (up to approximately 18 months)
Description: All adverse events, including serious adverse events, will be collected since the consent form is signed until 90th day after last administration of investigation products, either observed by investigator or by the spontaneous reported by subjects.
Arm/Group | Sintilimab+ Gemcitabine Plus Platinum | Placebo+Gemcitabine Plus Platinum
All-Cause Mortality (participants affected / at risk) | 65/179 | 71/178
Serious Adverse Events (participants affected / at risk) | 90/179 | 80/178
Other Adverse Events (participants affected / at risk) | 179/179 | 178/178
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sintilimab+ Gemcitabine Plus Platinum (N=179) | Placebo+Gemcitabine Plus Platinum (N=178)
Platelet count decreased (Investigations) | 32 | 32
White blood cell count decreased (Investigations) | 7 | 8
Neutrophil count decreased (Investigations) | 5 | 5
Amylase increased (Investigations) | 3 | 0
Lipase increased (Investigations) | 2 | 0
Pneumonia (Infections and infestations) | 22 | 14
Enteritis infectious (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 8 | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Immune-mediated pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Anaemia (Blood and lymphatic system disorders) | 6 | 6
Bone marrow failure (Blood and lymphatic system disorders) | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2
Pyrexia (General disorders) | 5 | 3
Asthenia (General disorders) | 2 | 0
Death (General disorders) | 2 | 5
Rash (Skin and subcutaneous tissue disorders) | 5 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 3
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 1 | 0
Platelet count increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 1
Sudden death (General disorders) | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 2
Hypochloraemia (Metabolism and nutrition disorders) | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 1 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 2
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Altered state of consciousness (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 2
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Speech disorder (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Immune-mediated endocrinopathy (Endocrine disorders) | 1 | 0
Hypophysitis (Endocrine disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 1 | 0
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Encephalitis (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sintilimab+ Gemcitabine Plus Platinum (N=179) | Placebo+Gemcitabine Plus Platinum (N=178)
White blood cell count decreased (Investigations) | 159 | 153
Neutrophil count decreased (Investigations) | 149 | 146
Platelet count decreased (Investigations) | 130 | 125
Aspartate aminotransferase increased (Investigations) | 43 | 35
Alanine aminotransferase increased (Investigations) | 42 | 44
Weight decreased (Investigations) | 35 | 24
Lymphocyte count decreased (Investigations) | 17 | 14
Blood creatinine increased (Investigations) | 16 | 13
Amylase increased (Investigations) | 14 | 6
Blood albumin decreased (Investigations) | 12 | 7
Blood glucose increased (Investigations) | 11 | 14
Gamma-glutamyltransferase increased (Investigations) | 10 | 12
Weight increased (Investigations) | 10 | 9
Blood bilirubin increased (Investigations) | 9 | 11
Anaemia (Blood and lymphatic system disorders) | 167 | 161
Nausea (Gastrointestinal disorders) | 71 | 73
Vomiting (Gastrointestinal disorders) | 58 | 61
Constipation (Gastrointestinal disorders) | 55 | 45
Diarrhoea (Gastrointestinal disorders) | 25 | 19
Abdominal distension (Gastrointestinal disorders) | 14 | 16
Decreased appetite (Metabolism and nutrition disorders) | 57 | 53
Hypophagia (Metabolism and nutrition disorders) | 28 | 15
Hypokalaemia (Metabolism and nutrition disorders) | 26 | 17
Hyponatraemia (Metabolism and nutrition disorders) | 26 | 33
Hypoalbuminaemia (Metabolism and nutrition disorders) | 25 | 21
Hypoproteinaemia (Metabolism and nutrition disorders) | 22 | 15
Hypocalcaemia (Metabolism and nutrition disorders) | 11 | 7
Hypochloraemia (Metabolism and nutrition disorders) | 9 | 13
Hyperglycaemia (Metabolism and nutrition disorders) | 8 | 13
Asthenia (General disorders) | 60 | 60
Pyrexia (General disorders) | 52 | 47
Chest discomfort (General disorders) | 13 | 10
Oedema peripheral (General disorders) | 9 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 27 | 22
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 19
Productive cough (Respiratory, thoracic and mediastinal disorders) | 9 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 12
Hiccups (Respiratory, thoracic and mediastinal disorders) | 6 | 9
Rash (Skin and subcutaneous tissue disorders) | 42 | 26
Pruritus (Skin and subcutaneous tissue disorders) | 22 | 10
Alopecia (Skin and subcutaneous tissue disorders) | 9 | 10
Pneumonia (Infections and infestations) | 40 | 28
Upper respiratory tract infection (Infections and infestations) | 13 | 11
Urinary tract infection (Infections and infestations) | 13 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 21
Ventricular extrasystoles (Cardiac disorders) | 10 | 3
Sinus tachycardia (Cardiac disorders) | 9 | 6
Supraventricular extrasystoles (Cardiac disorders) | 9 | 3
Hypothyroidism (Endocrine disorders) | 23 | 9
Hyperthyroidism (Endocrine disorders) | 10 | 6
Dizziness (Nervous system disorders) | 11 | 9
Headache (Nervous system disorders) | 10 | 7
Proteinuria (Renal and urinary disorders) | 21 | 15
Hepatic function abnormal (Hepatobiliary disorders) | 16 | 8
Insomnia (Psychiatric disorders) | 15 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-11-27): https://cdn.clinicaltrials.gov/large-docs/25/NCT03629925/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-17): https://cdn.clinicaltrials.gov/large-docs/25/NCT03629925/SAP_001.pdf